CLINICAL TRIAL: NCT02687607
Title: CLinical Assessment of WEB® Device in Ruptured aneurYSms
Brief Title: CLARYS: CLinical Assessment of WEB® Device in Ruptured aneurYSms
Acronym: CLARYS
Status: Completed | Type: Observational
Sponsor: Microvention-Terumo, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP15-001
Record Dates: First submitted 2016-02-16; First posted 2016-02-22 (Estimated); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Brain Aneurysm
Keywords: Endovascular; Brain aneurysm; Ruptured aneurysm
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm, Ruptured

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- WEB Aneurysm Embolization System: Subjects aged ≥ 18 years, but ≤ 80 years requiring treatment for single ruptured intracranial aneurysms.
  Interventions: Device: WEB Aneurysm Embolization System

INTERVENTIONS:
Device: WEB Aneurysm Embolization System

SUMMARY:
An observational non-randomized, multi-center, prospective assessment of the clinical utility of the WEB Aneurysm Embolization System in subjects with ruptured intracranial aneurysms deemed appropriate for endovascular treatment. The population being treated in this Registry is a subset of the CE marked indication.

DETAILED DESCRIPTION:
All eligible subjects presenting to the participating Registry Center will be considered for entry into the Registry. Up to 70 evaluable subjects meeting the Registry entry criteria will be enrolled.

An intermediary analysis will be performed when the first forty (40) subjects reaching the planned one month follow-up.

subjects will be followed per Institution's standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. The decision to use a WEB device to treat the patient has been made before and independently of the decision to include the patient in this Registry
2. Subject must be ≥ 18 years and < 80 years of age
3. Subject must have a single intracranial aneurysm ruptured within 30 days requiring treatment according to a multidisciplinary decision Definition: For the purposes of this study a ruptured IA patient is defined as a patient with computed tomography (CT), magnetic resonance imaging (MRI), or lumbar puncture (LP) evidence of subarachnoid hemorrhage attributed to the index aneurysm within the last 30 days.
4. If the subject has one or more additional aneurysm, the additional aneurysm must not require treatment in emergency or within 30 days of the index procedure
5. Subject with Hunt & Hess Score of I, II or III
6. Conventional or Flat-panel CT is performed within 6hrs prior to femoral puncture (or just before WEB placement if any clinical worsening is noted before the treatment) to assess absence of re-bleeding prior the treatment
7. Aneurysm to be treated must have the following characteristics i. Morphology - saccular ii. Location

   * Basilar apex (BA), or
   * Middle cerebral artery (MCA) bifurcation, or
   * Internal carotid artery (ICA) terminus, or
   * Anterior communicating artery (ACom), or
   * Anterior cerebral Artery (ACA), or
   * Posterior Communicating (PCom) iii. Diameter and height of the aneurysm is appropriate size for treatment with the WEB Aneurysm Embolization System per device Instructions for Use: Max width diameter 10mm iv. Aneurysm is a priori intended to be treated only with WEB
8. Subject must be considered by the physician to be available for subsequent visits
9. Subject must be able to comply with all aspects of the screening, evaluation, treatment, and the post-procedure follow-up schedule
10. Subject, or its legal representative, must have received information regarding the data collection and data protection within this clinical evaluation, or must have signed the informed consent when locally mandatory.

Exclusion Criteria:

1. Subject is greater than 80 years of age
2. Subject has a Hunt & Hess Score of IV or V
3. Subject has more than one aneurysm requiring treatment within 30 days of index procedure
4. Maximum aneurysm width is >10mm
5. Subject is female and pregnant or breast-feeding
6. Subject has a known coagulopathy
7. Subject has a known hemoglobinopathy or thrombocytopathy
8. Subject has lesion with characteristics unsuitable for endovascular treatment
9. Subject has vessel, tortuosity or morphology which could preclude safe access and support during treatment with clinical evaluation device
10. Subject has physical, neurologic or psychiatric conditions, which preclude Subject's ability to comply with all aspects of the screening, evaluation, treatment, and the post-procedure follow-up schedule
11. Subject has known hypersensitivity, which can not be treated, to any component of the clinical evaluation device, procedural materials, or medications commonly used during the procedure
12. Subject has received any investigational device for treatment of the target intracranial aneurysm prior to entry into this trial
13. Subject has an acute life-threatening illness other than the neurological disease to be treated in this trial
14. Subject has a life expectancy of less than 1 year due to other illness or condition (in addition to an intracranial aneurysm) Imaging Exclusion criteria
15. An additional aneurysm need to be treated during the index procedure
16. Microcatheter cannot reach Subject's aneurysm to allow necessary access to treat with WEB.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The decision to use a WEB device to treat the patient has been made before and independently of the decision to include the patient in this Registry
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-01; Primary Completion 2017-10-10 (Actual); Study Completion 2018-12-04 (Actual)

PRIMARY OUTCOMES:
Re-Bleed rate after treatment | 1 month
  Re-bleeding rate after treatment of the target aneurysm with WEB, during the period extending from post-procedure up to 1 month.
  Definitions:
  1. Re-bleeding from target aneurysm is defined as patent evidence of hemorrhage on CT or MRI AND hemorrhage is depicted in the same territory as the initial bleeding AND hemorrhage has increased in size compare to initial pre-operative CT
  2. Screening for re-bleeding: During hospital stay of the patient and up to 1-month, any worsening of the clinical status should lead to perform a non-enhanced CT or MRI.
  Or, as per-center standard care, non-enhanced CT or MRI might be performed systematically during hospital course.

SECONDARY OUTCOMES:
Aneurysm occlusion | 12 months
  Angiographic (conventional or CT-Angio or MR-Angio) occlusion at 12month based on WEB occlusion scale (WOS)

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Spelle, MD, PhD, Principal Investigator — CHU Bicetre
Locations (1):
- Service de Neuroradiologie, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CLinical Assessment of WEB device in Ruptured aneurYSms (CLARYS): 12-month angiographic results of a multicenter study — https://jnis.bmj.com/content/early/2022/07/26/neurintsurg-2022-018749
- See also: CLinical Assessment of WEB device in Ruptured aneurYSms (CLARYS): results of 1-month and 1-year assessment of rebleeding protection and clinical safety in a multicenter study — https://jnis.bmj.com/content/14/8/807